CLINICAL TRIAL: NCT05879640
Title: Sleep Disturbances for Children After Critical Care: Pilot Sleep Education Intervention
Brief Title: Sleep After Pediatric Critical Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Cydni Williams, Associate Professor, Oregon Health and Science University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 23234
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Pediatric; Critical Illness; Sleep Disturbance
MeSH Terms: conditions — Critical Illness; Parasomnias

STUDY DESIGN:
Intervention Model Description: Before-after
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Before- standard care (No Intervention)
- After- intervention (Other): Patients studied in this arm receive the new educational intervention delivered in conjunction with standard care
  Interventions: Behavioral: Sleep education

INTERVENTIONS:
Behavioral: Sleep education — Participants receive a handout about age appropriate sleep goals and tips for improving sleep. The handout also contains links to educational videos about sleep hygiene and the importance of sleep to healing after illness. The handout is reviewed with a clinician at bedside prior to hospital discharge.
  Arms: After- intervention

SUMMARY:
This study tests a pilot educational sleep intervention for children after critical care hospitalization.

DETAILED DESCRIPTION:
The investigators are conducting a before-after study evaluating an educational intervention delivered during hospitalization on sleep outcomes 1month after critical care hospitalization for children aged 6 to 18 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 years to 18 years inclusive
* Inpatient consult to Pediatric Critical Care and Neurotrauma Recovery Program

Exclusion Criteria:

* Abusive trauma
* Child protective services custody
* Prisoners
* Pregnancy
* Non-English speaking caregivers

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Sleep Disturbances Scale for Children | 1-month
  26-item parent report sleep measure; generates total T-score and 6 subscale T-scores (range 0-100, M 50, SD 10)

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory Scale (PedsQL) | 1-month
  Parent rated quality of life measure, age based; Generates total score 0-100

CONTACTS AND LOCATIONS:
Overall Officials: Cydni Williams, MD, MCR, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No